

Approved by the Nemours IRB: Valid from: 04/04/2014 through 04/03/2015

IRB# JAX: 332965

Abbreviated Study Title: LASST RPA Ancillary

### ADOLESCENT ASSENT FORM FOR YOUTH AGES 12-17

Your parent has given permission for you to be in a project called a research study. But first, we want to tell you all about it so you can decide if you want to be in it. If you don't understand, please ask questions. You can choose to be in the study, not be in the study or take more time to decide.

## What is the name of the study?

Long-Acting Beta Agonist Step Down Study (LASST) – Ancillary Study "Assessment of the Research Consent Process"

# Who is in charge of the study?

The doctor in charge of the study is Kathryn Blake, PharmD.

### What is the study about?

We know that it is sometimes difficult to understand all the medical information a doctor may give to you when you are at a doctor's appointment. We are trying to find better ways of communicating with children about medical information. We would like to find out how well you understand the information given to you about the study called "Long-Acting Beta Agonist Step Down Study".

## Why are you asking me to be in this study?

You are being asked to be in the study because you are interested in being in the study called "Long-Acting Beta Agonist Step Down Study".

### What will happen to me in the study?

At today's visit, we will have you read over the form that explains the "Long-Acting Beta Agonist Step Down Study". Then you and the study staff will sit in a room with your parent, and the study staff will ask you questions about the "Long-Acting Beta Agonist Step Down Study". You will have lots of chances to ask your questions about the study too. We will be audio recording your conversations with the study staff. This part will take about 15 minutes. After this part is over, we will ask you to look at some health information and then ask you a few questions about that information. This part will take about 3 to 5 minutes.

If you decide to be in the "Long-Acting Beta Agonist Step Down Study" you will do the same questions with the study nurse again at Visit 6. We will audio record it then too. The same parent who is with you at this visit will need to come with you at Visit 6. This will help us understand how well the study staff tells you about the study while you have been in it.

There is no benefit to you for being in this study. There are no risks for you being in this study either.

# Will I be paid to be in this study?

You will receive a \$10 Walmart gift card at this visit and Visit 6 for participating in this audiorecording of the communication between you and the study staff. There is additional payment if you participate in the main study, "Long-Acting Beta Agonist Step Down Study" which is described in the documents for that study.



Approved by the Nemours IRB: Valid for

Valid from: 04/04/2014

through 04/03/2015

IRB# JAX: 332965



Abbreviated Study Title: LASST RPA Ancillary

# Do I have to be in the study?

You don't have to do the study if you don't want to. If you are in the study, you can stop being in it at any time. Nobody will be upset with you if you don't want to be in the study or if you want to stop being in the study. The doctors and nurses will take care of you as they have in the past. If you have any questions or don't like what is happening, please tell the doctor or nurse.

You have had the study explained to you. You have been given a chance to ask questions. By writing your name below, you are saying that you want to be in the study.

Adolescent's Signature

Date

Name of Person Obtaining Assent

Signature of Person Obtaining Assent

Date